CLINICAL TRIAL: NCT03654222
Title: The Long-term Success of Cardiovascular Surgery in Takayasu Arteritis. 30 Years of Experience in Mexico, Beyond Forefront Techniques
Brief Title: The Long-term Success of Cardiovascular Surgery in Takayasu Arteritis
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Maria Elena Soto, MsC and PhD, RESEARCH DOCTOR, Instituto Nacional de Cardiologia Ignacio Chavez
Other Study IDs: 20142018
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Arteritis, Takayasu
MeSH Terms: conditions — Takayasu Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Cardiac surgery: Direct procedures in heart
- Organ preservation: Mainly renal autograft
- Bypass: Revascularization of affected organs or segments with Woven Dacron graft
- Exclusion: Resection of an affected organ (nephrectomy)
- Replacement: Replacement of affected aortic segment with a Woven Dacron graft
- Other: Any surgery that does not include the previous ones

SUMMARY:
Takayasu Arteritis (TA) affects medium and large caliber arteries causing stenosis, occlusion or aneurysms. It has great predilection for the aortic arch, subclavian and extracranial arteries. The global prevalence is of 1 to 2% per million inhabitants, which varies by geographical region. The main cause of death in TA is of cardiovascular origin and includes ischemic cardiomyopathy and valvular disease. The aim of this study was to evaluate the surgical experience according to the type of surgery in subjects with TA with and without inflammatory activity.

Methods: This was a retrospective, descriptive, cross-sectional study run between 1977 and 2017. Patients with Takayasu arteritis with more than 3 classification criteria according to the American College of Rheumatology (ACR) were included. The surgeries were classified as: Organ preservation, cardiac, bypass, exclusion and replacement. Inflammatory activity was evaluated.

DETAILED DESCRIPTION:
A review of the clinical records of patients diagnosed with TA with more than 3 criteria of the American College of Rheumatology (ACR) and undergoing some surgical procedure by the Surgery Service of the National Institute of Cardiology "Ignacio Chávez", in a period of time comprised between 1977 and 2016 was done. Patients of any gender and age who had been operated on by a surgical procedure registered in their medical record were included. Patients intervened in other institutions were excluded. The surgical event was classified into 6 groups: 1) organ-preservation surgery (mainly renal autograft); 2) Bypass (revascularization of affected organs or segments with Woven Dacron graft); 3) Replacement (replacement of affected aortic segment with a Woven Dacron graft); 4) Cardiac Surgery (direct procedures in heart); 5) Exclusion (resection of an affected organ (nephrectomy)), and 6) Other.

Inflammatory activity was evaluated according to the Dabague-Reyes criteria, in which a score greater than or equal to 5 is considered as active inflammation (9).

Statistical analysis: Variables with a loss of the sample data greater than 20% were excluded. The categorical variables were described by percentages and prevalences and the comparison were done by chi square or Fisher's exact test. A statistically significant level was considered when an error α <0.05 was found. Parametric numerical variables are described by measures of central tendency and the comparison is made by Student's T test. The survival analysis was performed using Kaplan-Meier. Ethical aspects were considered according to the Helsinky declaration.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any gender regardless of age that has a diagnosis of TA established by a rheumatologist,
* Have a surgical procedure registered in your medical record

Exclusion Criteria:

* Not having a digital, physical or microfilmed medical record
* Surgical procedures performed at another institution

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A review of clinical records of patients with diagnosis of Takayasu arteritis and undergoing some surgical procedure by the surgery service of the National Institute of Cardiology "Ignacio Chávez", in a period between 1977 and 2016 was conducted.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 1977-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Long-term survival rate surgery event | 45 years
  Observed in our study in relation to the mortality associated with the surgical event
Long-term survival according from other causes | 30 years
  According to the type of surgery in relation to mortality from other causes

SECONDARY OUTCOMES:
Arterial lesions | 30 years
  According to Numano's classification
Inflammatory activity | 30 years
  Evaluated according to the Dabague-Reyes criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Nacional Institute of Cardiology, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serra R, Butrico L, Fugetto F, Chibireva MD, Malva A, De Caridi G, Massara M, Barbetta A, Cannistra M, de Franciscis S. Updates in Pathophysiology, Diagnosis and Management of Takayasu Arteritis. Ann Vasc Surg. 2016 Aug;35:210-25. doi: 10.1016/j.avsg.2016.02.011. Epub 2016 May 27. PMID 27238990
- [Background] Hoffman GS. Takayasu arteritis: lessons from the American National Institutes of Health experience. Int J Cardiol. 1996 Aug;54 Suppl:S99-102. doi: 10.1016/s0167-5273(96)88778-x. PMID 9119532
- [Background] Lazzarin P, Pasero G, Marson P, Cecchetto A, Zanchin G. [Takayasu's arteritis. A concise review and some observations on a putative case reported by Giovanni Battista Morgagni (1761)]. Reumatismo. 2005 Dec;57(4):305-13. doi: 10.4081/reumatismo.2005.305. Italian. PMID 16380760
- [Background] SHIMIZU K, SANO K. Pulseless disease. J Neuropathol Clin Neurol. 1951 Jan;1(1):37-47. No abstract available. PMID 24538949
- [Background] Sharma BK, Jain S, Suri S, Numano F. Diagnostic criteria for Takayasu arteritis. Int J Cardiol. 1996 Aug;54 Suppl:S141-7. doi: 10.1016/s0167-5273(96)88783-3. PMID 9119516
- [Background] Park SJ, Kim HJ, Park H, Hann HJ, Kim KH, Han S, Kim Y, Ahn HS. Corrigendum to "Incidence, prevalence, mortality and causes of death in Takayasu Arteritis in Korea - A nationwide, population-based study" [Int. J. Cardiol., 235(2017), 100-104]. Int J Cardiol. 2017 Jul 1;238:182. doi: 10.1016/j.ijcard.2017.04.013. Epub 2017 Apr 24. No abstract available. PMID 28449826
- [Background] Dabague J, Reyes PA. Takayasu arteritis in Mexico: a 38-year clinical perspective through literature review. Int J Cardiol. 1996 Aug;54 Suppl:S103-9. doi: 10.1016/s0167-5273(96)88779-1. PMID 9119510
- [Background] Soto ME, Espinola N, Flores-Suarez LF, Reyes PA. Takayasu arteritis: clinical features in 110 Mexican Mestizo patients and cardiovascular impact on survival and prognosis. Clin Exp Rheumatol. 2008 May-Jun;26(3 Suppl 49):S9-15. PMID 18799047
- [Background] Lupi-Herrera E, Sanchez-Torres G, Marcushamer J, Mispireta J, Horwitz S, Vela JE. Takayasu's arteritis. Clinical study of 107 cases. Am Heart J. 1977 Jan;93(1):94-103. doi: 10.1016/s0002-8703(77)80178-6. PMID 12655
- [Background] Schmidt J, Kermani TA, Bacani AK, Crowson CS, Cooper LT, Matteson EL, Warrington KJ. Diagnostic features, treatment, and outcomes of Takayasu arteritis in a US cohort of 126 patients. Mayo Clin Proc. 2013 Aug;88(8):822-30. doi: 10.1016/j.mayocp.2013.04.025. Epub 2013 Jul 10. PMID 23849994
- [Background] Nazareth R, Mason JC. Takayasu arteritis: severe consequences of delayed diagnosis. QJM. 2011 Sep;104(9):797-800. doi: 10.1093/qjmed/hcq193. Epub 2010 Oct 15. No abstract available. PMID 20952441
- [Background] Rosa Neto NS, Shinjo SK, Levy-Neto M, Pereira RMR. Vascular surgery: the main risk factor for mortality in 146 Takayasu arteritis patients. Rheumatol Int. 2017 Jul;37(7):1065-1073. doi: 10.1007/s00296-017-3656-y. Epub 2017 Feb 21. PMID 28224216
- [Background] Ogino H, Matsuda H, Minatoya K, Sasaki H, Tanaka H, Matsumura Y, Ishibashi-Ueda H, Kobayashi J, Yagihara T, Kitamura S. Overview of late outcome of medical and surgical treatment for Takayasu arteritis. Circulation. 2008 Dec 16;118(25):2738-47. doi: 10.1161/CIRCULATIONAHA.107.759589. No abstract available. PMID 19106398
- [Background] Ishikawa K. Natural history and classification of occlusive thromboaortopathy (Takayasu's disease). Circulation. 1978 Jan;57(1):27-35. doi: 10.1161/01.cir.57.1.27. PMID 21760
- [Background] Saadoun D, Lambert M, Mirault T, Resche-Rigon M, Koskas F, Cluzel P, Mignot C, Schoindre Y, Chiche L, Hatron PY, Emmerich J, Cacoub P. Retrospective analysis of surgery versus endovascular intervention in Takayasu arteritis: a multicenter experience. Circulation. 2012 Feb 14;125(6):813-9. doi: 10.1161/CIRCULATIONAHA.111.058032. Epub 2012 Jan 9. PMID 22230484
- [Background] Mwipatayi BP, Jeffery PC, Beningfield SJ, Matley PJ, Naidoo NG, Kalla AA, Kahn D. Takayasu arteritis: clinical features and management: report of 272 cases. ANZ J Surg. 2005 Mar;75(3):110-7. doi: 10.1111/j.1445-2197.2005.03312.x. PMID 15777385
- [Background] Kaku Y, Aomi S, Tomioka H, Yamazaki K. Surgery for aortic regurgitation and aortic root dilatation in Takayasu arteritis. Asian Cardiovasc Thorac Ann. 2015 Oct;23(8):901-6. doi: 10.1177/0218492315591291. Epub 2015 Jun 18. PMID 26089524
- [Background] Miyata T, Sato O, Koyama H, Shigematsu H, Tada Y. Long-term survival after surgical treatment of patients with Takayasu's arteritis. Circulation. 2003 Sep 23;108(12):1474-80. doi: 10.1161/01.CIR.0000089089.42153.5E. Epub 2003 Sep 2. PMID 12952846
- [Background] Li J, Zhu M, Li M, Zheng W, Zhao J, Tian X, Zeng X. Cause of death in Chinese Takayasu arteritis patients. Medicine (Baltimore). 2016 Jul;95(27):e4069. doi: 10.1097/MD.0000000000004069. PMID 27399093
- [Background] Chiche L, Kieffer E, Sabatier J, Colau A, Koskas F, Bahnini A. Renal autotransplantation for vascular disease: late outcome according to etiology. J Vasc Surg. 2003 Feb;37(2):353-61. doi: 10.1067/mva.2003.84. PMID 12563206
- [Result] Carlson JA. The histological assessment of cutaneous vasculitis. Histopathology. 2010 Jan;56(1):3-23. doi: 10.1111/j.1365-2559.2009.03443.x. PMID 20055902